CLINICAL TRIAL: NCT02206880
Title: Examining DELIRIUM in Postoperative Cardiac Surgery Patient in Canada: Providing a National "Snapshot" of an Increasingly Devastating Complication
Brief Title: The Delirium-CS Canada Study
Acronym: DELIRIUM-CS
Status: Completed | Type: Observational
Sponsor: St. Boniface Hospital (Other)
Collaborators: Foothills Medical Centre (Other); Mazankowski Alberta Heart Institute (Unknown); London Health Sciences Centre (Other); Southlake Regional Health Centre (Other); Toronto General Hospital (Other); Hamilton Health Sciences Corporation (Other); Ottawa Heart Institute Research Corporation (Other); Royal Victoria Hospital, Canada (Other); Montreal Heart Institute (Other); New Brunswick Heart Centre (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Rakesh C. Arora, Principal Investigator, St. Boniface Hospital
Other Study IDs: DELIRIUM CS-Canada
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Delirium
Keywords: Thoracic Surgery; Delirium; Cardiopulmonary Bypass; Intensive Care
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Delirium is a prevalent complication following cardiac surgery that is under-recognized using current methods of delirium detection and that may be better identified through a systematic and standardized perioperative screening protocol.

The purpose of this study is to determine the incidence of postoperative delirium in the current era of cardiac surgery using a validated delirium-screening tool.

DETAILED DESCRIPTION:
Delirium is an acute confusional state characterized by fluctuating mental status, inattention, and either disorganized thinking or altered level of consciousness. It has long been recognized as a complication of cardiac surgery, a condition more likely to be experienced among elderly patients and those with greater comorbid disease burden. In recent years, increasing attention has been paid to the negative effect of delirium on post-operative outcomes, including long-term survival, freedom from hospital readmission and reduced cognitive and functional recovery. Despite this, little is still known about the true incidence of delirium following cardiac surgery, with published rates of delirium post-cardiac surgery ranging widely from 3% - 78%.

From September 1, 2014 to November 30, 2014, ALL patients undergoing cardiac surgery at each of the participating centers will be screened for post-operative delirium. Patients will NOT be excluded on the basis of urgency or procedure type. Delirium screening will be conducted for either up to 7 days following their date of surgery or up until their date of initial discharge from the intensive care unit, whichever comes first. Each center will be allowed to employ the delirium-screening tool currently in use at their institution provided that the tool is either the Intensive Care Delirium Screening Checklist (ICDSC) or Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). It is intended that either ICDSC or CAM-ICU, paired with a Richmond Agitation and Sedation Scale (RASS) or the Riker Sedation and Agitation Scale (SAS) be administered once per shift (i.e. with first assessment in the morning and a second assessment with the beginning of the evening shift). In addition, data regarding baseline demographic and clinical characteristics will be collected as well as data regarding the procedure performed (see Case Report Form (CRF). Patients will be considered as having had post-operative delirium if the results of at least one of the screening tests administered yielded a positive finding of delirium. In addition to reporting an overall rate of delirium, unadjusted and adjusted incidence rates of delirium will be reported by institution and for the entire cohort. Risk-adjustment will be performed using multivariate regression modeling techniques.

This study will be the first to report on incidence rates of delirium following cardiac surgery across multiple centers employing standardized screening methodologies. The results of this study will provide valuable insight into the true burden of delirium among patients having undergone a cardiac surgical procedure in the current era. This is the first step in creating a multifaceted delirium prevention/treatment clinical pathway for the cardiac surgery patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing cardiac surgery who are admitted to an ICU or CSRU following their procedure

Exclusion Criteria:

* Patients in whom delirium cannot be reliably identified (e.g., previous debilitating stroke, cerebral palsy, severe dementia, severe hearing disabilities or inability to understand English or French, active seizure disorder or Child-Pugh class B or C cirrhosis)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing cardiac surgery who are admitted to an ICU or CSRU following their procedure at twelve Canadian tertiary cardiac surgery centers in which patients are managed post-operatively in an intensive care unit (ICU) or cardiac surgery recovery unit (CSRU)
Sampling Method: Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Delirium following Cardiac Surgery | Delirium screening will be conducted for either up to 7 days following their date of surgery or up until their date of initial discharge from the intensive care unit, whichever comes first.
  Each center will be allowed to employ the delirium-screening tool currently in use at their institution provided that the tool is either the Intensive Care Delirium Screening Checklist (ICDSC) or Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). It is intended that either ICDSC or CAM-ICU, paired with a Richmond Agitation and Sedation Scale (RASS) or the Riker Sedation and Agitation Scale (SAS) be administered once per shift (i.e. with first assessment in the morning and a second assessment with the beginning of the evening shift). In addition, data regarding baseline demographic and clinical characteristics will be collected as well as data regarding the procedure performed (see Case Report Form (CRF). Patients will be considered as having had post-operative delirium if the results of at least one of the screening tests administered yielded a positive finding of delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh C. Arora, MD, PhD, FRCSC, Principal Investigator — St. Boniface General Hospital - Cardiac Sciences
Locations (12):
- Canada (12):
  - Foothills Medical Centre, Calgary, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - New Brunswick Heart Centre, Saint John, New Brunswick
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Derived] DELIRIUM-CS Investigators*; Canadian Cardiovascular Critical Care Society Investigator Group and the Canadian Critical Care Trials Group. Incidence of delirium after cardiac surgery: protocol for the DELIRIUM-CS Canada cross-sectional cohort study. CMAJ Open. 2017 Jul 13;5(3):E565-E569. doi: 10.9778/cmajo.20160136. PMID 28743102